CLINICAL TRIAL: NCT04871542
Title: Immune Checkpoint Inhibitor Toxicity (I-CHECKIT): A Prospective Observational Study
Brief Title: Immune Checkpoint Inhibitor Toxicity Risk Prediction in Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S2013; NCI-2021-01262 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2013 (Other: SWOG); SWOG-S2013 (Other: DCP); S2013 (Other: CTEP); UG1CA189974 (NIH)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, plasma, buffy coat
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, questionnaire): Patients undergo collection of a tissue sample at the start of their routine cancer treatment. Patients complete questionnaires at the start of cancer treatment, weeks 4, 12, 24, and 52. Patients will have the option of providing blood samples at several time points during the study.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood sample
  Other Names: Biological Sample Collection
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study examines how certain risk factors (such as age, gender, other medical conditions, and the type of immunotherapy used to treat the cancer) affect whether a patient with a malignant solid tumor will develop mild or serious side effects from the immunotherapy medications. Immunotherapy is the type of treatment that helps the body's immune system fight cancer. In the future, this information may help doctors make better decisions about cancer treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To both develop and independently validate a risk prediction model for Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher non-hematological immune-related adverse events (irAEs) in the first year of immune checkpoint inhibitor (ICI)-based therapy for the treatment of solid tumors.

SECONDARY OBJECTIVES:

I. To prospectively assess the incidence of any grade of non-hematological irAEs and grade 4 hematological irAEs on ICI-based therapy.

II. To observe the trajectory of patient-reported quality of life and health preferences over 12 months.

III. To observe the trajectory of patient-reported adverse events over 12 months using serial assessment with select Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) measures.

IV. To measure the burden of chronic, grade 1 and 2 toxicities using methods such as toxicity over time (ToxT).

V. To track patterns of treatment of irAEs and patterns of toxicity resolution.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To evaluate the cytokine toxicity (CYTOX) score, a composite measure derived from 11 different cytokine levels, both prior to ICI-based therapy and after 1 cycle of ICI-based therapy as a predictive signature for the development of irAEs.

II. To establish a repository of archival tissue and blood/serum specimens for potential predictive and/or prognostic markers of irAE risk.

ADDITIONAL OBJECTIVE:

I. To assess the feasibility of using electronic (e)PRO in a multi-center clinical trial setting.

OUTLINE:

Patients undergo collection of a tissue sample at the start of their routine cancer treatment. Patients complete questionnaires at the start of cancer treatment, weeks 4, 12, 24, and 52. Patients will have the option of providing blood samples at several time points during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be planning to receive ICI-based therapy for a solid tumor malignancy. This therapy must be given according to Food and Drug Administration (FDA) label or National Comprehensive Cancer Network (NCCN) guidelines at Category 1 or 2A and not in the context of a clinical trial
* Participants who have received prior ICI-based therapy must have completed ICI based therapy at least 180 days prior to registration
* Participants must not have discontinued any prior ICI-based therapy (if applicable) because of irAE
* Participants must not have received chemotherapy, biologic, or targeted-therapy within 21 days prior to registration
* Participants must have recovered from side effects of prior therapy to the following standards per treating physician's discretion:

  * =< Grade 1 for any non-hematologic side effects (excluding neuropathy and alopecia); lab-related parameters of liver and renal function will be considered at the discretion of the treating physician)
  * =< Grade 2 for neuropathy and/or alopecia
  * Grade 3 or less for any hematologic side effects
* Participants must be planning to begin standard of care ICI-based therapy within 3 calendar days after registration
* Participants must not be planning to receive ICI-based therapy in combination with chemotherapy or any other non-ICI therapy for treatment of their cancer
* Participants must be at least 18 years of age
* Participants must complete their history and physical examination within 28 days prior to registration
* Participants who can complete the S2013 Feasibility Questionnaire in English or Spanish must participate at the scheduled assessments
* Participants must be able to complete Patient-Reported Outcome (PRO) instruments in English, Spanish, or French and must be planning to complete PROs at all scheduled assessments
* Participants must complete the pre-registration (baseline) PRO forms within 14 days prior to registration
* Participants must be willing to participate in PRO data collection

  * Note: Prior to registration, participants must decide on their method (paper or electronic) of completing their follow-up questionnaires. Participants who elect electronic (ePRO) completion must have an iPhone, Android phone, or tablet with cellular or WiFi connectivity in order to download the Patient Cloud mobile applications onto the device (personal device or a site provisioned device for multi-users)
* Participants must be offered the opportunity to participate in the optional specimen banking
* Note: As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.

  * Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planning to receive ICI-based therapy for a solid tumor malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 2062 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-03-14 (Estimated)

PRIMARY OUTCOMES:
Occurrence of severe or worse non-hematological immune-related adverse event (irAE) | 52 weeks
  Adverse events will be recorded according to the physician rated Common Terminology Criteria for Adverse Events (CTCAE) scoring system.

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 | Baseline to 52 weeks
  PROMIS-29 Includes 4 questions to evaluate each of 7 domains (physical function, anxiety, depression, fatigue, sleep disturbance, social functioning, and pain interference) using a 5- point Likert scale, as well as a single item to assess pain severity on a 0-10 scale. The PROMIS-29 assesses severity levels of symptoms and their effect on the patient's functioning, assessed over the preceding 7-day period.
Change in PRO-CTCAE scores | Baseline to 52 weeks
  Patients report severity, frequency, and/or interference of toxicities. For this protocol the following 11 items will be assessed: fatigue interference, neuropathy severity and interference, nausea frequency and severity, shortness of breath severity and interference, presence of rash, itching severity, and diarrhea severity and interference over the preceding 7 days.
Change in PROMIS Cognitive Function- Short Form 4a version 2.0 scores | Baseline to 52 weeks
  Assesses patient-perceived cognitive deficits over the past 7 days. Facets include mental acuity, concentration, verbal and nonverbal memory, verbal fluency, and perceived changes in these cognitive functions. The extent to which cognitive impairments interfere with daily functioning, whether other people observe cognitive impairments, and the impact of cognitive dysfunction on quality of life are also assessed. The PROMIS Short Form Cognitive Function 4a is a questionnaire composed of 4 items rated on a 5 level scale, ranging from Never to Very often (Several times a day), with raw scores ranging from 5 to 20, with higher scores representing better cognitive function. In combination with the PROMIS-29, the use of this questionnaire allows the calculation of the PROMIS-Preference score, which quantifies the value participants place on different health states.
Change in toxicity over time (ToxT) | Baseline to 52 weeks
  ToxT is a collection of statistical codes in Statistical Analysis Software that generate plots depicting summary statistics or individual patient data over discrete timepoints, combined with longitudinal statistical analyses (repeated measures modelling, and time-to-event and AUC analyses).
Change in cytokine toxicity (CYTOX) score | Baseline to 1 cycle after ICI-therapy
  The relationship between the CYTOX score and the occurrence of irAE will be evaluated using area under the curve (AUC). Separate evaluations will be conducted using both cytokine levels determined both prior to ICI-based therapy and after 1 cycle of ICI-based therapy.

OTHER OUTCOMES:
Feasibility of the Patient Cloud electronic (e)PRO app | Up to 52 weeks
  Will be assessed by comparing the extent of missing data at each assessment time between participants choosing the Patient Cloud ePRO application (app) versus the use of paper forms. The participant experience of using the Patient Cloud ePRO app will also be assessed using a one-time questionnaire at the end of the participant's participation in the study

CONTACTS AND LOCATIONS:
Overall Officials: Krishna S Gunturu, Principal Investigator — SWOG Cancer Research Network
Locations (6):
- United States (6):
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa